CLINICAL TRIAL: NCT03027583
Title: The Effect of 6 Weeks Supplementation of Probiotic on Exercise-induced Intestinal Permeability in Trained Subjects - a Randomized, Double-blind, Placebo-controlled, Two Armed Parallel Group Trial.
Brief Title: The Effect of Probiotic Intervention on Intestinal Permeability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chr Hansen (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry); Signifikans ApS (Other)
Responsible Party: Sponsor
Organization: ChrHansen (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HND-GI-023
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Intestinal Permeability
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): 63 subjects will be randomized to the experimental arm. The experimental product is a vegetable capsule containing a probiotic strain. Subjects will consume 1-2 capsules daily together with breakfast, equivalent to a dose of 50 bill CFU for 6 weeks.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): 63 subjects will be randomized to the placebo arm.The placebo product is the same vegetable capsule as the experimental product, identical in composition, taste and appearance but without probiotics. Subjects will consume 1-2 capsules daily with breakfast for 6 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — 6 weeks daily oral intake of a probiotic strain.
  Arms: Probiotic
Dietary Supplement: Placebo — 6 weeks daily oral intake of placebo.
  Arms: Placebo

SUMMARY:
This trial is a single-site, randomised, double blind, placebo-controlled, two-armed parallel-group trial in healthy adult volunteers. The trial will investigate the effect of oral supplementation of a probiotic strain on the ability to attenuate exercise-induced deterioration of intestinal barrier function and gastrointestinal symptoms.

DETAILED DESCRIPTION:
The trial includes a run-in period of two weeks duration followed by a six weeks intervention period.

After having given their written informed consent, subjects will complete screening procedures to evaluate their eligibility for the trial and complete a run-in period of minimum two weeks duration to washout possible pre-trial probiotics. At the screening visit (visit 1), subjects will also perform a VO2max test on a running treadmill to determine their individual VO2max.

After baseline assessments at visit 2 and 3, the subjects will be randomly assigned to one of the two treatment groups (active or placebo product) in a ratio of 1:1. The two arms will be stratified for gender.

The subjects will consume 1-2 capsules once daily, together with breakfast, for six weeks starting at Day 1, the day after Visit 3. During the entire run-in and intervention period the subjects will be asked not to consume any other probiotic products. During the entire trial subjects should maintain their habitual life style in relation to physical activity level, diet and sleep habits.

At Visit 2, 3, 4 and 5, the small intestinal permeability will be evaluated by the L:R ratio measured in urine obtained 5 hours after oral ingestion of a lactulose and rhamnose solution. The permeability test will be performed in combination with a 1 hour treadmill running challenge when performed at Visit 3 and Visit 5. The treadmill run will be performed at a velocity corresponding to 80% of the subjects individually measured VO2max.

Faecal, urine and blood samples will be collected at Visit 2, 3, 4 and 5 for evaluation of the secondary objectives. The faecal samples collected will be: First bowel movement post-permeability test at Visit 2, first bowel movement post-exercise test at Visit 3, first bowel movement post-permeability test at Visit 4 and the first bowel movement post-exercise at Visit 5.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to any trial related procedures
2. Healthy (gastrointestinal symptoms are allowed, but not needed)
3. Weekly training load ≥ 4 hours within endurance sports as judged by the subject (minimum 1.5 hours of the training must be running activity)
4. Able to complete a 10 km run on a treadmill within 60 minutes, as judged by the subject
5. Willing to abstain from any probiotics products or medication known to alter gastrointestinal function throughout the participation of the trial

Exclusion Criteria:

1. Abdominal surgery which, as judged by the investigator, might affect the gastrointestinal function (except appendectomy and cholecystectomy)
2. Resting diastolic blood pressure ≥ 90 mmHg
3. Resting systolic blood pressure ≥ 140 mmHg
4. A current diagnosis of psychiatric disease
5. Systemic use of antibiotics, steroids (except contraceptives) or antimicrobial medication in the last 2 months
6. Daily usage of non-steroidal anti-inflammatory drugs in the last 2 months or incidental use in the last 2 weeks prior to screening
7. Usage of medications, except contraceptives, in the last 2 weeks prior to screening
8. Diagnosed inflammatory gastrointestinal disease
9. Lactose intolerance
10. Any other disease that, by the Investigators discretion, could interfere with the intestinal barrier function of the subject
11. Participation in other clinical trials in the past 2 months prior to screening
12. Regular use of probiotics in the last 2 months
13. Smoking and/or frequent use of other nicotine products
14. Desire and/or plans on changing current diet and/or exercise regime during the participation of this trial
15. Use of laxatives, anti-diarrheals, anti-cholinergics within last 2 months prior to screening
16. Use of immunosuppressant drugs within last 4 weeks prior to screening
17. Women: Pregnancy or lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 251 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Change in small intestine permeability | 6 weeks
  The effect of 6 oral supplementation of a probiotic strain versus placebo on small intestinal permeability measured as the change in urinary lactulose:rhamnose ratio following a 1 hour exercise challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Fergus Shanahan, Professor, Principal Investigator — Cork University Hospital
Locations (1):
- Atlantia Food Clinical trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Engel S, Mortensen B, Wellejus A, Vera-Jimenez N, Struve C, Brummer RJ, Damholt A, Woods T, Shanahan F. Safety of Bifidobacterium breve, Bif195, employing a human exercise-induced intestinal permeability model: a randomised, double-blinded, placebo-controlled, parallel group trial. Benef Microbes. 2022 Aug 3;13(3):243-252. doi: 10.3920/BM2021.0173. Epub 2022 Jul 22. PMID 35866597